CLINICAL TRIAL: NCT06249152
Title: A Pilot, Double-masked, Vehicle-controlled, Randomized Study to Evaluate the Safety and Tolerability of QLS-111 Versus Vehicle in Combination With Latanoprost Treatment in Subjects With Open-angle Glaucoma and/or Ocular Hypertension
Brief Title: Qlaris Study of QLS-111 in Combination With a PGA for OAG and/or OHT Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Qlaris Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QC-111-203; Apteryx (Other: Qlaris Bio, Inc.)
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Open-angle Glaucoma (OAG); Ocular Hypertension (OHT); Glaucoma
Keywords: Qlaris; OAG; Glaucoma; PGA therapy; Apteryx I; OHT; latanoprost
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma

STUDY DESIGN:
Intervention Model Description: Multi-site, double-masked, vehicle-controlled randomized prospective, parallel study of 14-day QPM dosing followed by 14-day BID dosing of QLS-111 (3 concentrations versus vehicle in combination with latanoprost. Dosing is OU.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study subjects, investigators, study staff, Sponsor and designates involved in the conduct, monitoring and outcome evaluation of the study will be masked to IP assignment identity until final database lock is complete. IP will be provided in in identical packaging. Unmasked statistician will prepare the randomization schedule.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental: QLS-111 ophthalmic solution (Experimental): Qlaris' IP, QLS-111 ophthalmic solution, provided in 3 concentrations (0.015%, 0.03%, and 0.075%), preservative free (PF), single-use units, masked.
  Interventions: Drug: QLS-111, 0.015%; Drug: QLS-111, 0.030%; Drug: QLS-111, 0.075%
- Placebo comparator: Vehicle ophthalmic solution (Placebo Comparator): Inactive control (0.00%), PF, single-use units, masked.
  Interventions: Drug: QLS-111 vehicle ophthalmic solution

INTERVENTIONS:
Drug: QLS-111, 0.015% — QLS-111 eyedrops applied QPM for 14 days the BID for 14 days.
  Other Names: QLS-111
  Arms: Experimental: QLS-111 ophthalmic solution
Drug: QLS-111, 0.030% — QLS-111 eyedrops applied QPM for 14 days the BID for 14 days.
  Other Names: QLS-111
  Arms: Experimental: QLS-111 ophthalmic solution
Drug: QLS-111, 0.075% — QLS-111 eyedrops applied QPM for 14 days the BID for 14 days.
  Other Names: QLS-111
  Arms: Experimental: QLS-111 ophthalmic solution
Drug: QLS-111 vehicle ophthalmic solution — Vehicle drops applied QPM for 14 days the BID for 14 days.
  Other Names: Vehicle; inactive control
  Arms: Placebo comparator: Vehicle ophthalmic solution

SUMMARY:
Qlaris Phase 2 clinical study investigating the safety, tolerability, and ocular hypotensive efficacy of QLS-111 in combination with latanoprost in open-angle glaucoma (OAG) and/or ocular hypertension (OHT) patients.

DETAILED DESCRIPTION:
Pilot, double-masked, vehicle-controlled, randomized, prospective parallel study of 14-day once daily evening (QPM) dosing, followed by 14-day twice daily (BID) dosing of an investigational product (IP), QLS-111, or vehicle as concomitant therapy with monotherapy latanoprost a PGA treatment that is administered QPM. Both eyes (OU) will be dosed. The study is comprised of seven (7) visits and approximately 28 days of IP dosing.

ELIGIBILITY:
Inclusion Criteria:

* 12 years or older
* Able and willing provide signed informed consent (assent)
* mild to moderate OAG or OHT in at least one eye and current or previous treatment with PGA. Exhibits decrease (i.e., >20% from reported pre- treatment) in intraocular pressure (IOP). Patient is willing to continue latanoprost throughout the study.
* IOP ≥19 mmHg at 08:00 hour (H) at qualification visits prior to randomization

Exclusion Criteria:

* History of active ocular disease other than mild to moderate OAG/OHT
* Nonresponse to and/or noncompliant with PGA treatment
* Use of other topical ocular medications with exception of the PGA which the patient will use throughout the study
* Moderate to severe glaucomatous damage in either eye
* Previous glaucoma intraocular surgery in either eye (e.g., trabeculectomy, tubes, cyclodestructive procedures, diode) with exception of selective laser trabeculoplasty (SLT) if done less than 12 months from screening, trabecular meshwork minimally invasive glaucoma surgery (MIGS) when combined with cataract surgery and done less than 12 months from screening.
* significant ocular trauma, or intraocular surgery (e.g., cataract extraction/intraocular lens insertion) or extensive retinal laser treatment, refractive surgery in either eye.
* Ocular infection, inflammation (e.g., uveitis), moderate to severe blepharitis/meibomitis and/or severe keratoconjunctivitis sicca in either eye at screening, history of herpes simplex keratitis, in either eye.
* Clinically significant retinal disease in either eye
* Clinically significant systemic or psychiatric disease
* Participation in any investigational study within 30 days prior to screening
* Pregnant or lactating

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-04-21 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Incidence of ocular treatment-emergent adverse events (TEAEs) | 28 days
  Ocular safety and tolerability
Clinically significant change in visual acuity | 28 days
  Ocular safety and tolerability
Clinically significant change in findings on slit lamp exam | 28 days
  Ocular safety and tolerability
Clinically significant change in findings on fundus exam | 28 days
  Ocular safety and tolerability
Incidence of systemic (TEAEs) | 28 days
  Systemic safety and tolerability
Clinically significant change in blood pressure | 28 days
  Systemic safety and tolerability
Clinically significant change in heart rate | 28 days
  Systemic safety and tolerability

SECONDARY OUTCOMES:
Change from baseline (CFB) of mean diurnal IOP in the study eye | 28 days
  Ocular hypotensive efficacy: diurnal IOP
CFB in IOP at various timepoints in the study eye | 28 days
  Ocular hypotensive efficacy: CFB for multiple timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Brandano, Study Director — Qlaris Bio, Inc.
Locations (1):
- Berkeley Eye Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Company website, pipeline — https://qlaris.bio